CLINICAL TRIAL: NCT03920020
Title: Comparison of The Effects of Concentric and Eccentric Isokinetic Exercises on Proprioception and Muscle Architecture in Patients With Knee Osteoarthritis
Brief Title: Comparison of The Effects of Concentric And Eccentric Isokinetic Exercises in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aysun Baki, principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA 17168
Record Dates: First submitted 2019-02-20; First posted 2019-04-18 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
Keywords: Concentric; Eccentric; Muscle Architecture; Proprioception
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the concentric isokinetic exercise group (Other): the concentric isokinetic exercise group will perform quadriceps and hamstring concentric isokinetic exercises in addition to the conventional physiotherapy and exercise program 3 times a week during 6 weeks.
  Interventions: Other: the concentric isokinetic exercise group; Other: the control group
- the eccentric isokinetic exercise group (Other): the eccentric isokinetic exercise group will perform quadriceps and hamstring eccentric isokinetic exercises in addition to the conventional physiotherapy and exercise program 3 times a week during 6 weeks.
  Interventions: Other: the eccentric isokinetic exercise group; Other: the control group
- the control group (Other): the control group will perform the standard exercise program predetermined by us consisting of stretching exercises and isometric strengthening (these exercises will be done at home, too) and the conventional physiotherapy program will be applied 3 times a week during 6 weeks.
  Interventions: Other: the control group

INTERVENTIONS:
Other: the concentric isokinetic exercise group — concentric isokinetic exercises
  Arms: the concentric isokinetic exercise group
Other: the eccentric isokinetic exercise group — eccentric isokinetic exercises
  Arms: the eccentric isokinetic exercise group
Other: the control group — conventional physiotherapy and standard therapeutic exercises predetermined by us

SUMMARY:
This study aims to compare the effects of concentric and eccentric isokinetic exercises on proprioception and muscle architecture in 42 patients with knee osteoarthritis enrolled the study.

DETAILED DESCRIPTION:
This study aims to compare the effects of concentric and eccentric isokinetic exercises on proprioception and muscle architecture in patients with knee osteoarthritis. 42 patients will be included in this study. Patients will be divided into three groups; concentric exercise group (n:14), eccentric exercise group (n:14) and control group (n:14). A conventional physiotherapy program and a standard therapeutic exercise program will be applied to all subjects. In addition to these exercise and physiotherapy programme, concentric and eccentric exercise groups will perform the exercises related to their groups. All three groups will participate in this program for a total of 18 sessions 3 times a week for 6 weeks. All groups will be subject to re-evaluation after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary knee osteoarthritis according to American College of Radiology
* Being radiographically K-L grade 2-3
* Presence of symptoms for at least 3 months
* Patients who have been planned a conventional physiotherapy programme because of knee osteoarthritis
* Presence of functional capacity for outpatient physical therapy

Exclusion Criteria:

* Patients with seconder knee osteoarthritis
* History of lower extremity or spine surgery
* History of intraarticular injection in last 1 month
* Patients with neurological disease that will affect muscle strength, balance and coordination

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Joint position sense | 6 weeks
  Joint position sense will be evaluated with isokinetic dynamometer at predetermined angles.
Ultrasonographic assessment of quadriceps and hamstring muscles | 6 weeks
  Ultrasonographic evaluation is an outcome measure to evaluate muscle structure. In our study ultrasonographic evaluation will be performed to determine the muscle structure (muscle thickness(mm), fascicle length(mm), pennation angle(degree)) of quadriceps and hamstring muscles. Muscle thickness will be defined as the distance between the deeper and upper aponeurosis. The pennation angle will be calculated as the angle of insertion of muscle fascicles into the deep aponeurosis. Fascicle length will be defined as the length of the fascicular path between the superficial and deep aponeurosis.

SECONDARY OUTCOMES:
WOMAC (Western Ontario & McMaster Universities Osteoarthritis Index) | 6 weeks
  WOMAC Osteoarthritis Index (score range 0-100) include 3 subscales and will be used to evaluate knee pain(score range 0-20), stiffness (score range 0-8), and functional limitation (score range -68). Womac is comprised of 24 items ( pain-5 items, stiffness-2 items, physical function-17 items). All items are scored on a scale of 0-4. Lower scores indicate lower disability.
Range of motion | 6 weeks
  Universal goniometer will be used for assessment of range of motion of the knee
Muscle strength assessment | 6 weeks
  isokinetic dynamometer test will be used.
Shortness of muscles assessment | 6 weeks
  universal goniometer will be used for assessment
Pain assessment: VAS (Visual analog scale) | 6 weeks
  VAS is used to measure the psycometric pain severity in some conditions and activities. A VAS is usually a 100 mm long horizontal line. The scale is most commonly anchored by "no pain" (line's left, score-0), "pain as bad as it could be" (line's right, score-100). the score is determined by measuring the distance between the "no pain" anchor and the patient's mark.
Balance assessment | 6 weeks
  Single leg standing test with eyes open and closed will be used. Timing is recorded.
The timed up and go test | 6 weeks
  TUG test is used to measure functional mobility. It gives an idea about patients walking ability, fall risk and balance. The patient is asked to get up, walk 3 meters and sit down again.Timing begins when the patient rise from the chair and stops when the patient sit down.
Sit to stand test | 6 weeks
  Patients stand up from and sit down on a chair as quickly as possible 5 times. Patients folded their arms across their chests. Timing is recorded.
Timed 10 meter walk test | 6 weeks
  This test is used to assess walking speed. Timing is recorded.
Short Form 12 (SF-12) health survey | 6 weeks
  SF-12 is an 12- item questionnare for assessing self-reported health related quality of life. It covers eight domains of health outcomes, including physical functioning, role physical, bodily pain, general health, vitality, social functioning,role-emotional, mental health. Sf-12 physical and mental component summary scales are scored. Lower SF-12 score indicated poorer physical and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Baki, phd student, Principal Investigator — Hacettepe University
Locations (1):
- Institute of Health Sciences, Ankara, Altındağ, Turkey (Türkiye)